CLINICAL TRIAL: NCT00370240
Title: Efficacy of Infiltration of Chlorhydrate of Ropivacaine in the Prevention of Chronic Breast Pain After Surgery for Breast Cancer.
Brief Title: Chlorhydrate of Ropivacaine and Breast Cancer Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: AstraZeneca (Industry); Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (CRH 05353A); EudraCT 2005-005691-32
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasms; Pain,Postoperative
Keywords: Female; Anesthetics,local
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ropivacaïne (Experimental)
  Interventions: Drug: Chlorhydrate de Ropivacaine
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Chlorhydrate de Ropivacaine — The Ropivacaïne group received 3mg/kg of 0.375% ropivacaïne(0.75% ropivacaïne, Astra, mixed with saline)
  Arms: Ropivacaïne
Other: placebo — The PCB group received saline solution in equal volume.
  Arms: placebo

SUMMARY:
The aim of the study is to evaluate the effect of local anesthetic (chlorhydrate of ropivacaine) to prevent chronic pain after breast surgery for cancer.

DETAILED DESCRIPTION:
An estimated 20-65% of women treated with breast surgery for breast cancer experience chronic pain in the treated breast. Patients will be randomize between: infiltration with chlorhydrate of ropivacaine at the time of breast surgery for cancer versus placebo.Intra-operative analgesia will be standardized as well as peri-operative pain management.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients treated by conservative surgery with axillary node dissection or treated by mastectomy with or without axillary node dissection or sentinel lymph node biopsy.
* ASA physical status 1, 2 or 3
* With a minimum life expectancy of 2 years
* Written informed consent

Exclusion Criteria:

* Any previous cancer other than breast cancer
* Allergies to local anesthesic and morphine
* Reported history of drug
* Pregnancy
* Homolateral breast surgery during the last 3 years
* Analgesic use pre-operatively
* Renal, pulmonary or liver major dysfunction
* Active malignant disease
* Unable to follow the protocol for any reason

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Comparing the frequencies of chronic breast pain 3 months after breast surgery evaluated by the Brief Pain Inventory in the two groups. | 3 months after surgery

SECONDARY OUTCOMES:
Visual Analogic Scale, Patient satisfaction with analgesic, consumption, neuropathic pain and depression/anxiety rating scale | 2 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aline H Albi-Feldzer, MD, Study Director — Centre René Huguenin - Saint-Cloud - France
Locations (1):
- René Huguenin Center, Saint-Cloud, France

REFERENCES:
- [Result] Albi-Feldzer A, Mouret-Fourme E E, Hamouda S, Motamed C, Dubois PY, Jouanneau L, Jayr C. A double-blind randomized trial of wound and intercostal space infiltration with ropivacaine during breast cancer surgery: effects on chronic postoperative pain. Anesthesiology. 2013 Feb;118(2):318-26. doi: 10.1097/ALN.0b013e31827d88d8. PMID 23340351